CLINICAL TRIAL: NCT03507543
Title: A Phase I, Open-label, Dose-escalation Study of the Safety and Pharmacokinetics of IMP4297 in Patients With Advanced Solid Tumors
Brief Title: The Safety and Pharmacokinetics of IMP4297 in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Impact Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMP4297-2016-AU01
Record Dates: First submitted 2018-01-08; First posted 2018-04-25 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Advanced Solid Tumours; Breast Cancer; Ovarian Cancer; Prostate Cancer; Primary Peritoneal Cancer
Keywords: Breast Cancer; Ovarian Cancer; Prostate Cancer; Advanced solid tumours; primary peritoneal Cancer
MeSH Terms: conditions — Breast Neoplasms; Ovarian Neoplasms; Prostatic Neoplasms | interventions — senaparib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IMP4297 (Experimental)
  Interventions: Drug: IMP4297

INTERVENTIONS:
Drug: IMP4297 — The dose levels will be escalated following a modified 3+3 dose escalation scheme.

SUMMARY:
This is a phase 1, First-In-Human, open label study, trialing a new PARP (poly-ADP ribose polymerase) inhibitor medication IMP4297 in participants with advanced solid tumour.

DETAILED DESCRIPTION:
This is a phase 1, First-In-Human, open label study, trialing a new PARP inhibitor medication IMP4297 in participants with advanced solid tumour.

Six different dosage cohorts 2mg, 6mg, 10mg, 20mg, 30mg and 40mg will be used to establish the maximum tolerated dosage. First participant in each dosing cohort will be administered one dose of IMP4297 capsule, followed by a wash out period of at least 5 half-lives or 7 days. Safety information such as pathology result or adverse events experienced will be collected following first dosing. This will be reviewed by the a safety review committee that is made up of the Principal Investigator, Medical Monitor, the study Sponsor and a representative from the Clinical Research Organisation, which will collectively determine if it is safe to proceed to continue with the next scheduled dosing cohort. Participant will proceed with repeat once daily dose at the same dose level for 3 weeks. Each repeat dose treatment cycle will be composed of 3 weeks (Day 1 to Day 21). IMP4297 will be administered by participants at home. Participants will be instructed to bring unused IMP4297 capsules with them to each visit for trial staff to review and confirm amount of IMP4297capsules taken since the last visit. The administration of the IMP4297 capsules will be recorded. Study drug compliance will be assessed using these records in conjunction with a count of unused IMP4297 capsules. Participants who are benefiting from IMP4297 may have the possibility of treatment beyond 1 year at the investigator's discretion. Participants who experience disease progression or unacceptable side effects, are not compliant with study protocol or in the opinion of the investigator will have IMP4297 administration discontinued and study participation will be terminated.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent Form
2. Age greater than or equal to 18 years
3. Histologically or cytologically documented, incurable, advanced solid malignancy that has progressed on, or failed to respond to, at least one prior systemic therapy
4. Evaluable or measurable disease per RECIST 1.1
5. ECOG performance status of 0 or 1
6. In the dose expansion stage, patients with BRCA (breast carcinoma) mutation will be enrolled. Patients with breast cancer, ovarian cancer and prostate cancer are preferred.

Exclusion Criteria:

1. Inadequate haematologic and organ function, defined by the following (haematologic parameters must be assessed greater than or equal to 14 days after a prior treatment, if any):

   1. Absolute neutrophil count <1500 cells/uL
   2. Haemoglobin <9 g/dL
   3. Total bilirubin >1.5 x the ULN, with documented liver metastases total bilirubin >3 x the ULN .
   4. AST and/or ALT >2.5 x the ULN, with documented liver metastases AST and/or ALT levels > 5 x the ULN.
   5. Serum creatinine > 1.5 x the ULN, or creatinine clearance < 50 mL/min based on a documented 24-hour urine collection.
   6. International normalized ratio (INR) > 1.5 x the ULN or activated partial thromboplastin time (aPTT) >1.5 x the ULN The INR applies only to patients who do not receive therapeutic anti-coagulation.
2. Any anti-cancer therapy, including chemotherapy, hormonal therapy, biologic therapy, radiotherapy within 4 weeks prior to initiation of study treatment with the following exceptions:

   1. Hormonal therapy with gonadotropin-releasing hormone (GnRH) agonists for prostate cancer
   2. Hormone-replacement therapy or oral contraceptives
   3. Palliative radiation to bone metastases > 2 weeks prior to Day 1
3. Adverse events from prior anti-cancer therapy that have not resolved to CTCAE Grade less than or equal to 1, except for alopecia
4. Clinical significant active infection
5. Known clinically significant history of liver disease, including viral or other hepatitis, current alcohol abuse, or cirrhosis
6. Known human immunodeficiency virus infection
7. New York Heart Association (NYHA) Class II or greater congestive heart failure; history of myocardial infarction or unstable angina within 6 months prior to Day 1; history of stroke or transient ischemic attack within 6 months prior to Day 1
8. Active or untreated brain metastasis
9. Pregnant (positive pregnancy test) or lactating women
10. Male or female patients of child-producing potential unwilling to use double barrier contraception: condoms, sponge, foams, jellies, diaphragm or intrauterine device (IUD), contraceptives (oral, injectable or parenteral), implanon, or other avoidance of pregnancy measures during the study and for 90 days after the last day of treatment
11. Inability to take oral medication, prior surgical procedures affecting absorption, or active peptic ulcer disease
12. Inability to comply with study and follow-up procedures
13. Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding that, in the investigator's opinion, gives reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or renders the patient at high risk from treatment complications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2017-02-03 (Actual); Primary Completion 2020-09-24 (Actual); Study Completion 2021-03-17 (Actual)

PRIMARY OUTCOMES:
The AEs (adverse event) of single and multiple doses of IMP4297 administered to participants with advanced solid tumors. | Each visit after IMP4297 administrated (through study completion, an average of 10 months)
  Evaluate the TEAE (treatment-emergent adverse event) of IMP4297
The maximum tolerated dose (MTD) and evaluate the dose limiting toxicities (DLTs) of IMP4297. | Within 28 days after IMP4297 administrated
  Evaluate DLT and determine the MTD

SECONDARY OUTCOMES:
Area Under Curve [AUClast, AUCINF and AUCtau] | Within 7 days after firstly single dose administrated
Area Under Curve [AUClast, AUCINF and AUCtau] | Within 16 days after first dose administrated in multiple dose cycle 1 (total 21 days in one cycle)
Maximum plasma concentration (Cmax) | Within 7 days after firstly single dose administrated
Maximum plasma concentration (Cmax) | Within 16 days after first dose administrated in multiple dose cycle 1 (total 21 days in one cycle)
Time at which Cmax occurred (Tmax) | Within 7 days after firstly single dose administrated
Time at which Cmax occurred (Tmax) | Within 16 days after first dose administrated in multiple dose cycle 1 (total 21 days in one cycle)
Trough Concentrations (Ctrough) | Within 7 days after firstly single dose administrated
Trough Concentrations (Ctrough) | Within 16 days after first dose administrated in multiple dose cycle 1 (total 21 days in one cycle)
Clearance (CL/F) | Within 7 days after firstly single dose administrated
Clearance (CL/F) | Within 16 days after first dose administrated in multiple dose cycle 1 (total 21 days in one cycle)
Volume of distribution (Vd/F) | Within 7 days after firstly single dose administrated
Volume of distribution (Vd/F) | Within 16 days after first dose administrated in multiple dose cycle 1 (total 21 days in one cycle)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Lickliter, Principal Investigator — Epworth Medical Centre; Paul Souza, Principal Investigator — St George Private Hospital
Locations (3):
- Australia (3):
  - Blacktown Hospital, Blacktown, New South Wales
  - St George Private Hospital, Kogarah, New South Wales
  - Nucleus Network, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gao B, Voskoboynik M, Cooper A, Wilkinson K, Hoon S, Hsieh CY, Cai S, Tian YE, Bao J, Ma N, Wang C, Zhang M, Li B, Guo M, Zhou R, Wang X, Xu C, de Souza P. A phase 1 dose-escalation study of the poly(ADP-ribose) polymerase inhibitor senaparib in Australian patients with advanced solid tumors. Cancer. 2023 Apr 1;129(7):1041-1050. doi: 10.1002/cncr.34662. Epub 2023 Jan 31. PMID 36718624